CLINICAL TRIAL: NCT04600661
Title: LOW LOAD RESISTANCE BLOOD FLOW RESTRICTION TRAINING VERSUS NEUROMUSCULAR TRAINING IN KNEE OSTEOARTHRITIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mai Mohamed Abdelkader Abdallah (Other)
Responsible Party: Sponsor-Investigator, Mai Mohamed Abdelkader Abdallah, Masters, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/002777
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: Blood flow restriction training
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Sixty Three patients of both genders with mild to moderate unilateral tibiofemoral OA, with age range from 45-60 years will be randomly assigned to 1 of 3 groups control group (Traditional therapy group) (n=21): patients will receive traditional training exercises (high load resistance training) Experimental group I (BFR training group) (n=21): patients will receive LLRT with BFR.
  Experimental group II (Neuromuscular training group) (n=21): patients will receive neuromuscular training exercises
Who Masked: Investigator, Outcomes Assessor
Masking Description: Sixty Three patients of both genders with mild to moderate unilateral tibiofemoral OA, with age range from 45-60 years will be randomly assigned to 1 of 3 groups using opaque, sealed envelopes, each containing the name of one of the groups. Each patient will sign an informed consent before starting the study (Appendix III). All patients will be referred by the orthopedic surgeon who will diagnose knee OA based on clinical and radiological examination. The investigator will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Traditional therapy group) (Experimental): control group (Traditional therapy group) (n=21): patients will receive traditional training exercises (high load resistance training
  Interventions: Other: Traditional exercise therapy
- Experimental group I (BFR training group) (Experimental): Experimental group I (BFR training group) (n=21): patients will receive LLRT with BFR.
  Interventions: Other: Traditional exercise therapy
- Experimental group II (Neuromuscular training group) (Experimental): Experimental group II (Neuromuscular training group) (n=21): patients will receive neuromuscular training exercises
  Interventions: Other: Traditional exercise therapy

INTERVENTIONS:
Other: Traditional exercise therapy — Neuromuscular training
  Other Names: Blood flow restriction training

SUMMARY:
This study will be conducted to compare the effect of BFR with LLRT versus neuromuscular training on quadriceps muscle strength, knee joint function and proprioception accuracy.

DETAILED DESCRIPTION:
PURPOSE:

This study will be conducted to compare the effect of BFR with LLRT versus neuromuscular training on quadriceps muscle strength, knee joint function and proprioception accuracy.

BACKGROUND:

Patients with knee OA may have reduction of tolerance of the high-load programs which is recommended for eliciting strength gains (Messier et al., 2013). Thus, for reducing disease risk and enhancing physical function, there is a need for effectively strengthening the quadriceps muscle while limiting pain and adverse joint loading in people with knee OA (Segal et al., 2015). Blood flow restriction (BFR) with low-load resistance training (LLRT) is an alternative to traditional strength training that can be used in knee OA with minimal adverse joint loading that is normally found in traditional strengthening programs(Pope et al., 2013). It is attained through applying pressure externally with a pneumatic cuff or tourniquet. The applied pressure occludes venous outflow while maintaining arterial inflow with intent to promote blood pooling in the capillary beds of the limb muscles distal to the tourniquet (Slysz et al., 2016). Kubota et al., (2008), showed that BFR can be applied during periods of immobilization to decrease disuse muscle atrophy of limbs. Also it can be combined with exercise which enhances muscular development. Resistance exercise appears to provide great muscular gains when combined with BFR (Slysz et al., 2016).

HYPOTHESES:

1. There will not be a significant difference between traditional training, BFR with LLRT and neuromuscular training on improving quadriceps muscle strength using HHD in patients with unilateral knee OA.
2. There will not be a significant difference between traditional training, BFR with LLRT and neuromuscular training on improving knee joint function on WOMAC questionnaire in patients with unilateral knee OA.
3. There will not be a significant difference between traditional training, BFR with LLRT and neuromuscular training on improving knee joint proprioception in patients with unilateral knee OA.

RESEARCH QUESTION:

Does blood flow restriction with low load resistance training and neuromuscular training have a significant effect over traditional rehabilitation protocol (stretching and strengthening for hip and knee muscles) on quadriceps muscle strength, knee joint function and proprioception accuracy in patients with unilateral knee OA?

ELIGIBILITY:
Inclusion Criteria:

* Age range from 45-60 years (Segal et al., 2015).
* Walk with painful knee OA without assistive devices (Bryk et al., 2016).
* Mild to moderate unilateral OA grade II-III (K/L) (Bryk et al., 2016).
* BMI < 30 kg/m² (not being classified as obese) (Bryk et al., 2016).
* Never participated in resistance training in the 3 months prior to their appointment (Jan et al., 2008)

Exclusion Criteria:

* Severe knee OA (grade IV according to K/L classification).
* Bilateral knee OA.
* Congenital or acquired inflammatory, rheumatic or neurological (systemic or local) diseases involving the knee.
* Repeated treatment with steroids.
* Secondary knee OA.
* Received joint replacement surgery in either Knee or/and hip.
* Cardiovascular and neuromuscular disorders
* Diabetic patients
* Psychiatric disorders.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 3 months
  Hand-Held Dynamometer for measuring muscle strength

SECONDARY OUTCOMES:
Knee joint function | 3 months
  Western Ontario and McMaster Universities osteoarthritis index for an Arab population for assessing knee function

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bryk FF, Dos Reis AC, Fingerhut D, Araujo T, Schutzer M, Cury Rde P, Duarte A Jr, Fukuda TY. Exercises with partial vascular occlusion in patients with knee osteoarthritis: a randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2016 May;24(5):1580-6. doi: 10.1007/s00167-016-4064-7. Epub 2016 Mar 12. PMID 26971109